CLINICAL TRIAL: NCT06644118
Title: A Pilot Clinical Study of OL-101 Injection in Patients with Relapsed or Refractory Multiple Myeloma (RRMM)
Brief Title: A Study of OL-101 Injection in Patients with Relapsed or Refractory Multiple Myeloma (RRMM)
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Zhejiang University (Other)
Collaborators: Overland Therapeutics (Unknown)
Responsible Party: Principal Investigator, He Huang, Professor, Zhejiang University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OL-101-001
Record Dates: First submitted 2024-09-28; First posted 2024-10-16 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-11

CONDITIONS: Multiple Myeloma
Keywords: OL-101; Multiple myeloma; Phase 1; single arm
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- OL-101 infusion (Experimental): This arm provides CAR-T treatment at the dose the patient is assigned to.
  Interventions: Biological: OL-101 infusion

INTERVENTIONS:
Biological: OL-101 infusion — OL-101 infusion will be administered to patients via IV infusion at the assigned dose.

SUMMARY:
This clinical trial aims to characterize the safety of OL-101 and establish the recommended dose for future research and to evaluate the efficacy of OL-101 (Dose expansion).

DETAILED DESCRIPTION:
This study will evaluate the safety and efficacy of OL-101, a chimeric antigen receptor T cell (CAR-T) therapy directed against B-Cell Maturation Antigen (BCMA) and G Protein-Coupled Receptor Class C Group 5 Member D (GPRC5D). This study is a single-arm, open-label, early exploratory clinical trial, conducted in two phases: dose escalation and dose expansion in adults with multiple myeloma. The trial begins with the dose-escalation phase that focus on safety and tolerability, with interval assessments for potential dose escalation or de-escalation. Recommended dose will be selected at the completion of the dose escalation stage in the dose expansion stage. The study aims to assess safety, pharmacokinetic/pharmacodynamic profiles, and efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Documented diagnosis of multiple myeloma according to the 2014 IMWG diagnostic criteria
* Relapsed/refractory multiple myeloma as defined by:

  1) Received at least 3 prior lines of MM treatment (must include a PI, an IMiD, and an anti-CD38 antibody).

  2）Disease progression within 12 months of the most recent anti-MM therapy; or disease progression within the past 6 months and subsequently lack response to the most recent line of therapy.
* Measurable disease at screening as defined by any of the following:

  1. Serum monoclonal paraprotein (M-protein) level ≥1.0 g/dL or urine M-protein level ≥200 mg/24 hours; or
  2. Light chain multiple myeloma without measurable disease in the serum or the urine: Serum immunoglobulin free light chain ≥10 mg/dL and abnormal serum immunoglobulin kappa lambda free light chain ratio.
* Positive expression of either BCMA or GPRC5D on bone marrow plasma cells; must be GPRC5D expression positive if previously received BCMA targeted therapy
* ECOG 0-1
* Expected life expectancy exceeds 12 weeks
* Adequate bone marrow reserve or organ function meeting the following criteria:

  1. Hemoglobin ≥ 70 g/L
  2. Platelet count ≥ 50 × 10^9/L
  3. Absolute lymphocyte count ≥ 0.3×10^9/L
  4. Absolute neutrophil count ≥ 1.0 × 10^9/L
  5. Alanine aminotransferase (ALT) and Aspartate aminotransferase (AST) ≤ 2.5 times the upper limit of normal (ULN)
  6. Total bilirubin ≤ 2 times ULN; except in subjects with congenital bilirubinemia (such as Gilbert syndrome, in which case the direct bilirubin ≤1.5 × ULN is required)
  7. Creatinine clearance ≥ 60 mL/min (calculated by Cockcroft-Gault equation).
  8. corrected serum calcium ≤12.5 mg/dL (≤3.1 mmol/L) or free ionized calcium ≤6.5 mg/dl (≤1.6 mmol/L)
  9. SpO2>92% on room air
  10. Left ventricular ejection fraction (LVEF) ≥ 50% as assessed by echocardiogram; no clinically meaningful pericardial effusion by ultrasound

Exclusion Criteria:

* Solitary plasmacytoma
* Known active central nervous system (CNS) involvement or exhibits clinical signs of CNS involvement of multiple myeloma.
* Received allogeneic stem cell transplant; received autologous stem cell transplant within 12 weeks before screening
* Active second primary malignant tumor, exclude the following: cured non- melanoma skin cancer, non-metastatic prostate cancer, cervical carcinoma in situ, ductal or lobular carcinoma in situ of the breast
* Any other significant medical disease, abnormality, or condition that, in the investigator judgment, may make the patient unsuitable for participation in the study or put the patient at risk.
* Plasma cell leukemia, Waldenström's macroglobulinemia, POEMS syndrome, or primary AL amyloidosis.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2024-10-23 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLT) | Within 28 days post CAR-T infusion
  Adverse events will be assessed based on the CTCAE 5.0
Treatment emergent adverse event (TEAE) incidence and severity | From aphresis till 1 year after CAR-T infusion or start of a new anti-cancer therapy, whichever is earlier
  Adverse events will be assessed based on the CTCAE 5.0

SECONDARY OUTCOMES:
Level of Immunogenicity | Baseline until 2 years after CAR-T infusion or withdrawn from the study, whichever comes first
  To assess the presence of antibodies to OL-101 (ADA)
Level of RCL | Baseline until 2 years after CAR-T infusion or withdrawn from the study, whichever comes first
  To determine whether Replication Competent Lentivirus (RCL) is present in patient that receive OL-101
Overall response rate (ORR) | Baseline until 2 years after CAR-T infusion or withdrawn from the study, whichever comes first
  Proportion of subjects with PR or above
Minimal residual disease (MRD) negative rate | Baseline until 2 years after CAR-T infusion or withdrawn from the study, whichever comes first
  Proportion of subjects with MRD negative status as defined by the IMWG response criteria
Duration of response (DOR) | Baseline until 2 years after CAR-T infusion or withdrawn from the study, whichever comes first
  The time from the initial response to therapy until the disease progression or relapse.
Progression-free survival (PFS) | Baseline until 2 years after CAR-T infusion or withdrawn from the study, whichever comes first
  The time from CAR-T cell infusion to the first assessment of disease progression or death from any cause.
Overall survival (OS) | Baseline until 2 years after CAR-T infusion or withdrawn from the study, whichever comes first
  The time from CAR-T cell infusion to death from any cause.
Cmax of OL-101 | Baseline until 2 years after CAR-T infusion or withdrawn from the study, whichever comes first
  The maximum concentration of the CAR-T cells will be measured to assess OL-101 in vivo expansion and persistence.
Tmax of OL-101 | Baseline until 2 years after CAR-T infusion or withdrawn from the study, whichever comes first
  The time of the maximum concentration will be measured to assess OL-101 in vivo expansion and persistence.
AUC 0-28days of OL-101 | Baseline until 2 years after CAR-T infusion or withdrawn from the study, whichever comes first
  Area under the curve will be measured to assess OL-101 in vivo expansion and persistence.
Serum cytokines | Baseline until 2 years after CAR-T infusion or withdrawn from the study, whichever comes first
  The levels of cytokines will be measured, such as IL-6 and ferritin.
Serum soluble circulating BCMA (sBCMA) | Baseline until 2 years after CAR-T infusion or withdrawn from the study, whichever comes first
  Serum soluble circulating BCMA will be measured to explore its potential relationship to response or resistance.

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Beijing Gobroad Boren Hospital, Beijing, Beijing Municipality
  - The Affiliated Hospital of Northwest University Xi'an No.3 Hospital, Xi’an, Shanxi
  - The first affiliated hospital, College of Medicine, Zhejiang University, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No